CLINICAL TRIAL: NCT06140563
Title: Prospective Study of Micro-CT Imaging to Quantify Dialyzer Clotting in Patients With End Stage Kidney Disease Undergoing Hemodialysis
Brief Title: Variability in Micro-CT Imaging Results to Quantify Dialyzer Clotting
Acronym: ClotVar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0201
Record Dates: First submitted 2023-11-13; First posted 2023-11-20 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Hemodialysis Complication; Anticoagulants
Keywords: dialyzer fiber clotting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal anticoagulation dosing (Experimental): Patients are dialyzed during three consecutive hemodialysis sessions with an FX800 Cordiax dialyzer, blood flow of 300mL/min, dialysate flow of 500mL/min and ultrafiltration according to the needs of the patient. At the start of the dialysis session, the normal amount of anticoagulation is administered.
  Interventions: Other: anticoagulation dosing
- Reduced anticoagulation dosing (Experimental): Patients are dialyzed during three consecutive hemodialysis sessions with an FX800 Cordiax dialyzer, blood flow of 300mL/min, dialysate flow of 500mL/min and ultrafiltration according to the needs of the patient. At the start of the dialysis session, only one quarter of the normal amount of anticoagulation is administered.
  Interventions: Other: anticoagulation dosing

INTERVENTIONS:
Other: anticoagulation dosing — In one arm the normal amount of anticoagulation is administered at the dialysis start, while this is only a quarter of the normal amount of anticoagulation in the other arm.

SUMMARY:
Different cross-over studies have been performed investigating dialyzer fiber patency in different dialysis setups. Herewith, post dialysis micro computed tomography (CT) images of the dialyzer were compared. For the best interpretation of such results, one should have an idea about the intrapatient variability. There is also no clue about the impact of long distance transportation and long cold storage on the reproducibility of the micro CT images. Another bottle neck is that, up till now, no biochemical parameter or test has been found associated with the outcome of dialyzer fiber patency post dialysis.

The present study therefore aims at determining the intrapatient variability and the impact on the micro CT results of long distance transportation and long cold storage of the dialyzers. Also, whole blood thrombin generation tests are performed to look for associations with the micro CT results.

DETAILED DESCRIPTION:
During recent years, different coagulation studies were performed using micro computed tomography (CT) scanning of hemodialyzers post dialysis as a marker for fiber blocking. Each of these studies investigated the impact of either anticoagulation strategy, dialysis strategy, or hemodialyzer type in a cross-over study design in which each patient served as his/her own control.

To date, we still need to answer some remaining questions related to studies using micro CT before we can expand the research and clinical applications to a larger scale:

First, the power of such cross-over studies, with a single session per study arm, depends also partially on the variability over time in the micro CT results within a single patient. While the resolution (25µm) and reproducibility of the micro CT process is established, patients' coagulation status will cause the largest variability in dialyzer outcome among consecutive dialysis sessions, e.g. variation due to infection or vascular access problems. This type of intrapatient variability, quantifying dialyzer outcome with micro CT from comparable but different dialysis sessions, has not yet been studied. Evaluation of the inter- and intra-patient variability of micro CT of dialyzers in chronic hemodialysis patients will inform whether this novel method can be used as an endpoint in future interventional trials of novel anticoagulants.

Second, the micro CT imaging technique, recently paraphrased as the gold standard to quantify clotting, is a very valuable technique in research settings. Clinical practice would profit more from a less burdensome marker of hemodialyzer performance as measured during the dialysis session (not only at the end of a dialysis session). However, none of the available online dialysis machine parameters (i.e., transmembrane pressure, arterial and venous pressure, online clearance monitoring), nor visual scoring of the dialyzer or venous chamber, nor assessment of dialyzer mass post-treatment correlated well with the results of micro CT. Also, the commonly used biochemical parameters only focus on one aspect in the coagulation cascade or/and are not sensitive enough to measure variations in the coagulation system of the patient. As a consequence, they are poorly related to dialyzer outcome as quantified with micro CT. While thrombin generation (TG) is commonly determined in plasma to identify global coagulation phenotype, whole blood TG (WB-TG) tests better mimic physiology by involving also the intrinsic blood cells and platelets, making it a potential biomarker test for coagulation, and this requires investigation.

Third, the previously described studies were all executed at the Ghent University Hospital where dialyzers are prepared for scanning on the spot (i.e., rinsed, dried and stored at 5°C), and with only a short transport time (15min) from the clinic to the micro CT scanner. No hard evidence however exists whether dialyzers, after being prepared for micro CT in a different place, might be transported by flight in e.g. isolated boxes (lasting hours to days). This study will be conducted in collaboration with Regeneron (New York) where a subset of 10 dialyzers will be shipped, imaged using Regeneron's micro CT scanner, and shipped back to Ghent University for repeat imaging.

The main aims of the proposed study are therefore:

1. to determine intrapatient variability of dialyzer fiber blocking as measured by micro CT scanning
2. to investigate whether longer transportation of dialyzers might impact reproducibility of micro CT results by comparing micro CT results between long and short transportation times of dialyzers
3. to determine the anticoagulant effect size of low molecular weight heparin by evaluating the difference in dialyzer fiber patency between full dose and low dose (1/4 dose) low molecular weight heparin treatment, which will inform sample size determination for future interventional studies of other anticoagulants

ELIGIBILITY:
Inclusion Criteria:

* stable chronic hemodialysis patient
* well functioning vascular access

Exclusion Criteria:

* ultrafiltration rate higher than 4 litre per session
* use of antiplatelets or anticoagulants (apart from acetylsalicylic acid)
* known coagulation disorder
* active inflammation
* malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Intrapatient variability of dialyzer fiber patency | 2 months
  The intrapatient variability of the dialyzer fiber patency (i.e. percentage open fibers post dialysis) and the intraclass correlation coefficient (ICC) of fiber patency are calculated from the results of the post dialysis micro CT images of the dialyzer, as scanned after three consecutive dialysis sessions with the same anticoagulation dosing: one week with full anticoagulation and one week with reduced (1/4) anticoagulation.
  Outcome = intrapatient variability of the percentage open fibers. Tool = micro CT scanning and computer-based determination of fiber patency.

SECONDARY OUTCOMES:
Impact of dialyzer storage and transport on micro CT images of dialyzer fibers | 3 months
  After initial scanning of the 60 dialyzers, 10 of these dialyzers will be transported to Regeneron (New York), where they will be scanned with a local micro CT scanner. After sending them back to Ghent University Hospital, dialyzers will be re-scanned. In the meantime, 10 other dialyzers (out of the 60 dialyzers) will be stored, after initial scanning, in a fridge in Ghent University Hospital. They will be re-scanned together with the ten dialyzers coming back from Regeneron.
  From all these micro CT images, fiber patency will be derived and comparisons are made between the results before versus after transport, and before versus after longer storage in the fridge.
  Outcome = comparisons between the percentage open fibers in the same filter either being transported or stored.
  Tool = micro CT scanning and computer-based determination of fiber patency.
Association between whole blood thrombin generation test and fiber patency | 2 months
  During each dialysis session, blood is sampled at the dialysis start and end to perform a whole blood thrombin generation test. Post dialysis, dialyzers are scanned with a micro CT scanner and the corresponding fiber patency is derived.
  Outcome = Associations between parameters of the whole blood thrombin generation test and the dialyzer fiber patency.
  Tools = Whole blood thrombin generation tests on blood samples and micro CT scanning and computer-based determination of fiber patency.
Difference in fiber patency using normal versus reduced anticoagulation dosing. | 2 months
  Patients are followed three dialysis sessions per week, one week with full anticoagulation dosing and one week with reduced (1/4) anticoagulation dosing. Post dialysis, dialyzers are scanned with a micro CT scanner and the corresponding fiber patency is derived.
  Outcome = Comparisons between the percentage open fibers in dialyzers after a session with full anticoagulation versus after a session with reduced anticoagulation.
  Tool = micro CT scanning and computer-based determination of fiber patency.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No